CLINICAL TRIAL: NCT06092502
Title: The Effectiveness of Graded Motor Imagery Therapy Applied in Addition to the Traditional Physiotherapy Program in Shoulder Impingement Syndrome
Brief Title: Shoulder Impingement Syndrome and Graded Motor Imagery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nuray Alaca (Other)
Responsible Party: Sponsor-Investigator, Nuray Alaca, Assoc. Prof. Nuray Alaca, Head of Physiotherapy and Rehabilitation Department, Acibadem University
Organization: Acibadem University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATADEK-2023/11
Record Dates: First submitted 2023-10-13; First posted 2023-10-23 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Shoulder Pain; Shoulder Impingement Syndrome
Keywords: Shoulder Pain; graded motor imagery
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Physiotherapy Program (Active Comparator): This group included strengthening exercises will be applied, including various joint movements and strengthening exercises applied in physiotherapy clinics.
  Interventions: Other: Traditional Physiotherapy Program
- Traditional Physiotherapy Program and Graded Motor Imagery Therapy (Experimental): The three different treatment techniques include left/right discrimination training, explicit motor imagery exercises and mirror therapy. These techniques are delivered sequentially but require a flexible approach from the patient and clinician to move forwards, backward and sideways in the treatment process to suit the individual. With patience, persistence and often lots of hard work, GMI gives new hope for treatment outcomes.
  Interventions: Other: Graded Motor Imagery; Other: Traditional Physiotherapy Program

INTERVENTIONS:
Other: Graded Motor Imagery — The three different treatment techniques include left/right discrimination training, explicit motor imagery exercises and mirror therapy. These techniques are delivered sequentially but require a flexible approach from the patient and clinician to move forwards, backward and sideways in the treatment process to suit the individual. With patience, persistence and often lots of hard work, GMI gives new hope for treatment outcomes.
  Other Names: Traditional Physiotherapy Program
  Arms: Traditional Physiotherapy Program and Graded Motor Imagery Therapy
Other: Traditional Physiotherapy Program — This protocol included stretching and strengthening exercises

SUMMARY:
Graded motor imagery (GMI): used successfully in chronic, complex and painful clinical conditions accompanied by many pain and movement problems; It is a treatment, education and rehabilitation process that is based on recently obtained scientific data and current clinical studies, is individually adapted and approaches the individual holistically with a biopsychosocial model. Nowadays, it is frequently used in the treatment of some neurological diseases. In addition, these approaches are also used in the treatment of some orthopedic diseases including chronic pain. There are a limited number of studies in which the mentioned approaches are used together in stages, and the stages are mostly used alone. There is only one study in the literature on subacromial pain syndrome (SAS), which is the most common cause of shoulder pain and causes radiator cuff problems. Stage 2 SAS patients were included in the study and only one phase of GMI treatment was used in addition to the traditional physiotherapy program. Despite these positive results in favor of GMI, the fact that there is no study using the entire GMI treatment in SAS shows us that a randomized controlled and blinded study with high evidence value should be conducted on this subject. In addition, determining the effect of GMI on changes in central nervous system such as fear of pain, two-point discrimination, and left/right lateralization speed and accuracy task will help fill the literature gaps on this subject. In the light of this information, the question of planned master's thesis study is the effect of GMI treatment applied in addition to traditional physiotherapy in SAS on pain level, joint range of motion, functionality, pain-related fear, two-point discrimination and left/right lateralization speed and accuracy compared to only traditional physiotherapy. whether it is superior or not.

ELIGIBILITY:
Inclusion Criteria:

* 20-50 years of age with complaints of shoulder pain in the anterio-lateral region lasting more than 6 weeks, with a positive Neer impingement test and/or a positive Hawkins-Kennedy test
* Additionally, patients must have at least one of the symptoms listed. These symptoms are: painful arch on active shoulder elevation, pain with resisted shoulder external rotation in abduction at 90°, and a positive empty can test.

Exclusion Criteria:

* Having had a steroid injection into the shoulder within the last 3 months

  * Previous surgery on the neck, thoracic spine or shoulder
  * Red flags (e.g. tumor, fracture, metabolic diseases, rheumatoid arthritis, osteoporosis, resting blood pressure greater than 140/90 mmHg, history of long-term steroid use)
  * History of shoulder dislocation, subluxation, fracture, adhesive capsulitis, frozen shoulder, or cervical or thoracic surgery
  * History of full-thickness rotator cuff tear
  * History of cervical disc herniation in the last 6 weeks
  * History of breast cancer on the involved side
  * Isolated acromioclavicular joint pathology (i.e., pain directly localized over the acromioclavicular joint).
  * Signs of cervical radiculopathy, radiculitis, or referred pain originating from the cervical spine
  * Receiving treatment for shoulder pain in the last 3 months
  * Being currently pregnant (Dunning, 2022)
  * Scoring ≤24 on the Standardized Mini Mental Test was determined.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-12-13 (Estimated); Study Completion 2025-12-13 (Estimated)

PRIMARY OUTCOMES:
The Numerical Rating Scale (NPRS-11) | Change from baseline range of motion at 6th week
  The Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain.0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
The Shoulder Pain and Disability Index | Change from baseline score of The Shoulder Pain and Disability Index at 6th week
  The Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability between 0 to 100, with a higher value indicating worse condition.
Global Rating of Change scale (Patient Satisfaction) | Change from baseline Global Rating of Change scale at 6th week
  Patient satisfaction regarding improvement in shoulder function will be evaluated by the Global Rating of Change scale. All participants will be asked to rate their condition after a six-week intervention period compared to baseline by indicating whether they have improved significantly, improved slightly, unchanged, deteriorated slightly, or deteriorated significantly between -3 to +3, with a higher value indicating better condition in this study.
Central Sensitization Scale | Change from baseline score of Central Sensitization Scale scale at 6th week
  Central Sensitization Scale, which can be applied in the presence of chronic pain, is used in central sensitization syndromes. It consists of two parts. Part A of the scale includes a Likert scale (0-4 points) that questions health-related symptoms. This section is scored from 0 to 100, with higher numbers being associated with a higher degree of central sensitization. Scores of 40 and above indicate the presence of central sensitization. In section B, it questions whether any of the central sensitization syndromes have been diagnosed before.

SECONDARY OUTCOMES:
Range of motion | Change from baseline range of motion at 6th week
  Shoulder range of motion is the capability of a joint to go through its complete spectrum of movements.
Pressure Pain Threshold | Change from baseline Pressure Pain Threshold at 6th week
  A digital pressure algometer will be applied to the web space of the foot opposite the trigger point. Participants are instructed to say "stop" or "pain" so the stimulus can be terminated "when the sensation first transitions from pressure to pain" (pain threshold).
Pain Catastrophizing Scale | Change from baseline score of Pain Catastrophizing Scale at 6th week
  The Pain Catastrophizing Scale (PCS) is a 13-item self-report measure designed to assess catastrophic thinking related to pain among adults with or without chronic pain.The person may score a total of 52 (Pain Catastrophizing Scale). A high score indicates a high level of catastrophic.
Fear avoidance belief questionnaire (FABQ) | Change from baseline score of Fear avoidance belief questionnaire at 6th week
  Fear avoidance belief questionnaire FABQ) is a questionnaire based on the fear-avoidance model of exaggerated pain perception. The FABQ measures patient's fear of pain and consequent avoidance of physical activity (PA) because of their fear.There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs. There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24)
The two-point discrimination test | Change from baseline two-point discrimination at 6th week
  The two-point discrimination test is used to assess if the patient is able to identify two close points on a small area of skin, and how fine the ability to discriminate this are. It is a measure of tactile agnosia, or the inability to recognize these two points despite intact cutaneous sensation and proprioception.
Left/right discrimination (Lateralization) | Change from baseline Left/right discrimination at 6th week
  Right-Left Discrimination will be evaluated with Recognise™ applications (Shoulder and Hand) developed by the "Neuro Orthopedic Institute".
Kinesthetic and Visual Imagery Questionnaire (KVIQ) | Change from baseline Kinesthetic and Visual Imagery Questionnaire at 6th week
  Motor imagery ability will be assessed with the Kinesthetic and Visual Imagery Questionnaire (KVIQ). The participant gives a score between 1 and 5 for the image he/she imagines: "1 point: no image, 5 points: as clear as the original." This process is repeated for each task and at the end of the survey, kinesthetic imagery score, visual imagery score and total score are calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuray ALACA, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided